CLINICAL TRIAL: NCT05632250
Title: A Prospective, Multi Centre, Interventional, Non-comparator, Open Label Study to Demonstrate the Efficacy, Safety, and Performance of ConvaFoam™ Silicone, ConvaFoam™ Border and ConvaFoam™ Non-adhesive Dressings in the Management of Indicated Chronic Wound Types.
Brief Title: A Prospective, Multi Centre, Interventional, Non-comparator, Open Label Study to Demonstrate the Efficacy, Safety, and Performance of ConvaFoam™ Dressings in the Management of Indicated Chronic Wound Types.
Acronym: MORGEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WC-22-427
Record Dates: First submitted 2022-11-09; First posted 2022-11-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Chronic Ulcer of Leg or Foot; Pressure Injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Post Market Clinical Follow Up Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ConvaFoam dressings (Other): All participants wounds will be assessed and allocated a dressing based upon the investigator's clinical judgement. They will receive either ConvaFoam Border, Silicone or Non-Adhesive for up to 12 weeks as part of their standard of care
  Interventions: Device: ConvaFoam

INTERVENTIONS:
Device: ConvaFoam — ConvaFoam™ Border, ConvaFoam™ Non-Adhesive, and ConvaFoam™ Silicone dressings are designed to provide a moist wound healing environment. These dressings are designed to manage excess exudate levels which may further damage the wound bed and surrounding skin. Patient's wounds will be assessed and a dressing from the above will be applied as part of their normal standard of care. The wounds will be assessed on a weekly basis for up to 12 weeks.
  Other Names: ConvaFoam Silicone; ConvaFoam Border; ConvaFoam Non Adhesive

SUMMARY:
A prospective, multi centre, interventional, non-comparator, open label study to demonstrate the efficacy, safety, and performance of ConvaFoam™ dressings in the management of indicated chronic wound types.

DETAILED DESCRIPTION:
A prospective, multi centre, interventional, non-comparator, open label study to demonstrate the efficacy, safety, and performance of ConvaFoam™ Silicone, ConvaFoam™ Border and ConvaFoam™ Non-Adhesive dressings in the management of Chronic leg ulcers (including diabetic foot ulcers) and Pressure Injuries (Grade II and above)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over
* Patients able and willing to provide informed consent
* Patients with wounds with a duration of no less than 2 months and no more than 12 months
* Patients must be willing to complete the QoL (quality of life) questionnaires via a valid email address
* Patients with at least one, but no more than two of the same wound indications which would require dressing according to the stage of the wound:

  * Chronic ulcers (Venous, arterial, mixed aetiology or diabetic foot ulcers)
  * Pressure Injury Stage II or greater
* Patients must be willing to attend visits as per schedule in protocol

Exclusion Criteria:

* Patients with known allergies to any of the materials used in the dressing
* Patients with known malignant wounds
* Patients requiring any oxidising agents such as hydrogen peroxide or hypochlorite solutions
* Patients, who in the opinion of the Investigator, are considered as unsuitable for any other reason
* Patients with chronic conditions such as autoimmune disorders in an acute flare phase, which in the opinion of the investigator would directly impact wound healing, use of immunosuppressant medications may be allowed if they have been on a stable dose and regimen over the past three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
To measure efficacy of ConvaFoam dressings in the exudate management of chronic wounds. | 12 weeks
  This will be measured by:
  Lack of strike through
  Loss of edge seal/adherence,
  Dressing leakage/seepage
  Dislodgement
  Need for dressing change

SECONDARY OUTCOMES:
To measure the performance of ConvaFoam dressings when used to manage chronic wound progression as per the instructions for use | 12 weeks
  Performance will be measured by documenting the progress of the wound through a weekly standard wound assessment where progression with be measured by changes to the wound healing status from deteriorating to static, static to improvement or improved to healed
To measure the performance of ConvaFoam dressings from a care health Care Practitioners Practitioners Perspective when used in accordance with the instructions for use | 12 weeks
  As part of the study schedule Health Care Professionals to complete a questionnaire at the end of study to assess:
  Ease of use
  Ease of removal ( Atraumatic)
  Wear time (meets recommended guidelines in IFU)
To measure the performance of ConvaFoam dressings in the management of chronic wounds from a patient perspective when used in accordance with the instructions for use | 12 weeks
  As part of the study schedule patients will be asked to complete a quality of life questionnaire on their first and final visit to measure:
  Dressing comfort ( patient satisfied with dressing comfort and able to resume activities of daily living
To measure the safety of Convafoam dressings when used to manage chronic wounds in accordance with the instructions for use | 12 weeks
  Any device related adverse events such as wound complications, maceration, blistering, breakdown of peri wound skin edges or changes to skin integrity will be documented and reported as per protocol
To measure the safety of Convafoam dressings when used to manage chronic wounds in accordance with the instructions for use | 12 weeks
  Any device related adverse events such will be documented and reported as per protocol

CONTACTS AND LOCATIONS:
Overall Officials: Kerem Ozere, MD, Study Director — Medical Director
Locations (5):
- United States (5):
  - Foot and Ankle Specialists of the Mid-Atlantic, Hagerstown, Maryland
  - NYU Langone Health, Mineola, New York
  - Foot and Ankle Specialsts of the Mid-Atlantic, Raleigh, North Carolina
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Hope Vascularity & Podiatry, PLLC, Houston, Texas

IPD SHARING:
Plan to Share IPD: No